CLINICAL TRIAL: NCT02382133
Title: Comparison of Nasal and Forehead Oximetry in Critically Ill Patients at Risk for Decreased Peripheral Perfusion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Lynn Schallom, Research Scientist, Washington University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 201408123
Record Dates: First submitted 2015-02-10; First posted 2015-03-06 (Estimated); Results first posted 2017-06-07 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-05

CONDITIONS: Hypotension; Pressure Ulcer
MeSH Terms: conditions — Hypotension; Pressure Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nasal alar oxygen sensor (Other): Application of a nasal alar oxygen sensor
  Interventions: Device: Nasal alar oxygen sensor

INTERVENTIONS:
Device: Nasal alar oxygen sensor — Application of a nasal alar oxygen sensor

SUMMARY:
Continuous pulse oximetry monitoring is the standard of care in critically ill patients in emergency departments, operating rooms and intensive care units. In patients with poor peripheral perfusion (low blood flow) due to peripheral vascular disease, low body temperature, or shock and the use of medications to raise the blood pressure, clinicians have difficulty obtaining an accurate measurement. This study compares the accuracy of forehead oximetry sensors to nasal alar sensors to lab oximetry measures and on the rate of device related pressure ulcers with both.

DETAILED DESCRIPTION:
Continuous pulse oximetry monitoring is the standard of care in critically ill patients in emergency departments, operating rooms and intensive care units. In patients with poor peripheral perfusion (low blood flow) due to peripheral vascular disease, low body temperature, or shock and the use of medications to raise the blood pressure, clinicians have difficulty obtaining an accurate measurement. Several studies have demonstrated the utility of forehead sensor measurements under these clinical conditions. Forehead sensor measurement is considered to be a more central measurement than with digit or ear sensors. However the sensor requires a head band for accurate measurement. On a regular basis, the forehead sensor has led to pressure ulcer development at Barnes-Jewish Hospital despite following vendor recommendations for alternating placement every 8 hours from one side of the forehead to the other. An alternate sensor placed on the nose has recently demonstrated rapid detection of induced drops in oxygen saturation. It has also demonstrated correlation with arterial oxygen saturation measured in a clinical laboratory. The oxygen saturation measurement from the nose is also considered a central measurement. However, studies of the nose sensor were conducted in healthy subjects or during anesthesia care over several hours. Therefore, research is needed to examine the accuracy of the nose sensor in the ICU patient population. In addition, due to concerns for sensor related pressure ulcers in patients with decreased perfusion, the sensor needs to be evaluated for extended periods of time.

ELIGIBILITY:
Inclusion Criteria:

1. Presence of an existing arterial catheter for blood sampling and one of the following:

1. Difficulty obtaining a consistent signal from a digit or ear sensor or
2. On pressors of at least 0 .10 mcg/kg/min of norepinephrine or
3. Core temperature < or equal to 35 degrees C

Exclusion Criteria:

1. Anatomic impediments (burns, wounds, dressings, etc.) to placement of the sensor on the forehead or nasal alar
2. History of known dyshemoglobinemias evidenced by carboxyhemoglobin levels > 10% or methemoglobin level > 2%
3. Severe anemia with hemoglobin < 5 g/dL
4. Pregnant women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2014-10; Primary Completion 2016-07 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marilyn E Schallom, RN, PhD, Principal Investigator — Barnes-Jewish Hospital at Washington University
Locations (1):
- Barnes-Jewish Hospital at Washington University, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schallom M, Prentice D, Sona C, Arroyo C, Mazuski J. Comparison of nasal and forehead oximetry accuracy and pressure injury in critically ill patients. Heart Lung. 2018 Mar-Apr;47(2):93-99. doi: 10.1016/j.hrtlng.2017.12.002. PMID 29402444

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Nasal Alar Oxygen Sensor
Started | 43
Completed | 10
Not Completed | 33
Not completed — Death | 22
Not completed — transfer out of ICU | 4
Not completed — Physician Decision | 2
Not completed — arterial catheter loss | 4
Not completed — pressure injury both sites | 1

BASELINE CHARACTERISTICS:
Arm/Group | Nasal Alar Oxygen Sensor
Number analyzed (Participants) | 43
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 24
  >=65 years | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.1 (16.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26
  Male | 17
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 43

OUTCOME MEASURES:

1. Primary Outcome: Accuracy as Indicated by Co-oximetry Measure of Arterial Oxygen Saturation
Description: accuracy of sensor measure was defined as sensor measurements within 3% of co-oximetry measures
Time Frame: 24 hours
Population: Nasal sensor unable to obtain a signal 7% of measures on enrollment, Forehead sensor unable to obtain signal 32% of measures on enrollment.
Measure: Count of Participants; unit: Participants
Arm/Group | Nasal Alar Oxygen Sensor
Number analyzed (Participants) | 43
Participants | 43

2. Secondary Outcome: Device Related Pressure Ulcer
Description: assessment for development of pressure ulcer at forehead sensor, "OxiMaxTM, Nellcor,Covidien" and nasal alar sensor, "Alar One-SenseTM, Xhale Assurance"
Time Frame: 5 days
Population: incidence of any pressure injury
Measure: Number; unit: participants
Arm/Group | Nasal Alar Oxygen Sensor
Number analyzed (Participants) | 43
participants | 2
Statistical Analysis 1: Comparison: Nasal Alar Oxygen Sensor; Test type: Superiority — comparing nasal and forehead oximetry sensor pressure ulcer incidence; p = .006, Chi-squared

ADVERSE EVENTS:
Arm/Group | Nasal Alar Oxygen Sensor
All-Cause Mortality (participants affected / at risk) | 22/43
Serious Adverse Events (participants affected / at risk) | 0/43
Other Adverse Events (participants affected / at risk) | 0/43

LIMITATIONS AND CAVEATS:
50% the patients expired after being placed on comfort care prior to final collection

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No